CLINICAL TRIAL: NCT05035199
Title: Spiritual Resources and Distress in Patients With Affective Disorders
Status: Completed | Type: Observational
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02859
Record Dates: First submitted 2021-07-15; First posted 2021-09-05 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Mood Disorders
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with psychiatric disorders: Patients with psychiatric disorders of the affective spectrum.
  Interventions: Behavioral: Spiritual Distress and Resources Questionnaire (SDRQ)

INTERVENTIONS:
Behavioral: Spiritual Distress and Resources Questionnaire (SDRQ) — The SDRQ is a validated self-rating instrument to assess spiritual distress and resources. It focuses on beliefs, attitudes, experiences and practices of various kinds (every day and extraordinary), as well as on (dis-)connectedness. It consists of 22 items covering three subscales: spiritual resources, spiritual distress, and spiritual coping (Peng-Keller et. al., 2020, submitted). We constructed five additional questions to find out more why patients want to include spiritual aspects in their treatment.

SUMMARY:
In this study, the investigators want to assess spiritual resources, spiritual distress and spiritual coping in patients with psychiatric disorders of the affective spectrum with a new designed questionnaire the Spiritual Distress and Resources Questionnaire (SDRQ)

DETAILED DESCRIPTION:
The inclusion of the spiritual dimension in healthcare has been a recommendation of the World Health Organization (WHO) since 1984. According to the WHO, 'spiritual' refers "to those aspects of human life relating to experiences that transcend sensory phenomena. This is not the same as 'religious', though for many people the spiritual dimension of their lives includes a religious component. The spiritual aspect of human life may be viewed as an integrating element holding together the physical, psychological and social dimensions. It is often perceived as being concerned with meaning and purpose". Today there is a growing body of scientific evidence for therapeutic relevance of the spiritual dimension in different fields of medical health care. Based on this increasing scientific evidence, medical associations such as the Royal College of Psychiatrists recommend the assessment of spiritual needs for therapeutic goals. Despite those long-standing calls and findings, these recommendations have not yet been widely implemented. Even in palliative care, patients indicate that their spiritual concerns are often inadequately addressed. Many clinicians report that they lack the required communication skills to adequately address spiritual concerns, while patients are not used to bring up their spiritual needs by themselves. As spiritual needs can only be integrated into care delivery if known to the practitioners, an explicit assessment is necessary. There are numerous instruments to assess spiritual aspects in the context of health care research - but only few to be used in a clinical context. Furthermore, there are many instruments that take into account the specific spiritual needs at the end of life in palliative care, while there are fewer established instruments in the care of chronic diseases. To close this gap, the investigators constructed and validated a new screening tool for assessing spiritual distress and resources, the Spiritual Distress and Resources Questionnaire (SDRQ) in patients with chronic pain in a previous project within the National Research Program "Smarter Health Care" (NRP 74).

The results of this NRP 74 project showed clearly: Spiritual aspects are considered as important in the context of chronic pain by health care professionals and patients alike. They could be important resources to be integrated in a multimodal pain therapy.

In this study, the investigators want to assess spiritual resources, spiritual distress and spiritual coping in patients with psychiatric disorders of the affective spectrum. To compare the results with the results of chronic pain patients, similar questionnaires as in the above mentioned study within NRP 74 will be used. Additionally, the investigators want to assess the proportion and characteristics of patients who wish spiritual aspects to be integrated in the therapeutic setting. Overall, the goal is to create knowledge to adequately address spiritual aspects in those patients who wish the integration of their spiritual needs into treatment.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Sufficient command of German language as assessed by local study coordinator
* Psychiatric disorder of the affective spectrum (depressive disorder, anxiety disorder, obsessive-compulsive disorder, adjustment disorder, somatoform disorder)

Exclusion Criteria:

* Cognitive disorders that would impair participation in assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To investigate the objectives, 220 psychiatric patients suffering from an affective disorder (ICD F3/F4) will be recruited consecutively. Because we assess a questionnaire with 22 items for our primary objective, the number of 220 patients seems reasonable. The project population consists of psychiatric patients at the outpatient and day-clinics of the Center for Social Psychiatry, Department of Psychiatry, Psychotherapy and Psychosomatics, University Hospital for Psychiatry of Zurich.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Spiritual distress, spiritual resources and spiritual coping as assessed with the SDRQ | 6 months
  To what extent do psychiatric patients with disorders of the affective spectrum have spiritual distress, spiritual resources and spiritual coping strategies?
Characteristics of patients as assessed with the sociodemographic questionnaire | 6 months
  What characterizes patients who want spirituality to be included in their treatment in comparison to patients who do not want this?
Comparison of the results of the SDRQ with the results of chronic pain patients | 6 months
  Are the results specific to patients with disorders of the affective spectrum in comparison to patients with chronic pain?

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rufer, Prof. Dr., Principal Investigator — PUK Zürich
Locations (1):
- PUK Zürich, Zurich, Switzerland

REFERENCES:
- [Background] World Health Organization (1985) Handbook of Resolutions and Decisions of the World Health Assembly and the Executive Board Vol. II 1973-1984. Geneva.
- [Background] WHO Expert Committee on Cancer Pain Relief and Active Supportive Care & World Health Organization. (1990). Cancer pain relief and palliative care. Report of a WHO expert committee [meeting held in Geneva from 3 to 10 July 1989]. World Health Organization. https://apps.who.int/iris/handle/10665/39524
- [Background] Bussing A, Baumann K, Hvidt NC, Koenig HG, Puchalski CM, Swinton J. Spirituality and health. Evid Based Complement Alternat Med. 2014;2014:682817. doi: 10.1155/2014/682817. Epub 2014 Jan 30. No abstract available. PMID 24616739
- [Background] Gerbershagen K, Trojan M, Kuhn J, Limmroth V, Bewermeyer H. [Significance of health-related quality of life and religiosity for the acceptance of chronic pain]. Schmerz. 2008 Oct;22(5):586-93. doi: 10.1007/s00482-008-0656-6. German. PMID 18478272